CLINICAL TRIAL: NCT06165757
Title: The Effects of Non Harmonic and White Noise on Human Pain Sensitivity: a Study of Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Noise and pain sensitivit
Record Dates: First submitted 2023-11-09; First posted 2023-12-11 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-10

CONDITIONS: Pain
Keywords: Noise; Pain
MeSH Terms: conditions — Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- noise on pain (Experimental): Comparison of pain sensitivity before and after hearing noise among 15 subjects in each group.
  Interventions: Behavioral: noise stimulation

INTERVENTIONS:
Behavioral: noise stimulation — Apply non harmonic and white noise sound stimuli to the subjects, and then measure the threshold and tolerance values of pressure pain, cold pain, and electrical pain.

SUMMARY:
Study the effects of 60dB and 80dB white noise, 50-70dB and 70-90dB non harmonic tones on the basic pain threshold of subjects, including the threshold and tolerance of electrical stimulation pain,the threshold and tolerance of cold pain stimulation, and the threshold and tolerance of tenderness stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 35, regardless of gender
* No serious chronic diseases
* There is no self-reported history of chronic opioid drug use or neuropathy

Exclusion Criteria:

* A history of alcohol or drug abuse
* Pregnant or lactating
* Severe cardiovascular, kidney, or liver diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
mechanical pain sensitivity | from the study beginning to 30 min after the procedure
  Each participant was measured using the pressure pain threshold and tolerance (tested by a pressure meter), which lower value present higher pain sensitivity
cold pain sensitivity | from the study beginning to 30 min after the procedure
  Each participant was measured using the cold pain threshold and tolerance (tested by immersion the hand in 4℃ water), which lower value present higher pain sensitivity
electrical pain sensitivity | from the study beginning to 30 min after the procedure
  Each participant was measured using the cold pain threshold and tolerance (tested by a electrical stimulator), which lower value present higher pain sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes